CLINICAL TRIAL: NCT04404582
Title: Analysis of the Clinical Characteristics for the Critical Ill Patients With Klebsiella Pneumoniae Infection: A Multi-center Research in the Intensive Care Units
Brief Title: Clinical Characteristics for the Critical Ill Patients With Klebsiella Pneumoniae Infection
Status: Completed | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, associate senior doctor, Fujian Provincial Hospital
Other Study IDs: K2019-06-031
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Drug Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Klebsiella pneumoniae: patients with Klebsiella pneumoniae infection had different results of the drug sensitivity test. we compared the prognosis of these patients.

SUMMARY:
The detection of Klebsiella pneumoniae virulence gene and antibiotics resistance gene takes a long time and high cost with equipment requirements. Distinguishing the Klebsiella pneumoniae by gene were late for clinical treatment. Therefore, the investigators aim to study the clinical characteristics of critically ill patients with Klebsiella pneumoniae infection which expressed different drug sensitivity test results.

DETAILED DESCRIPTION:
Clinical data of adult patients in integrated ICUs of 6 hospitals of Fujian Province China from January 2015 to July 2019 were collected, who had been examined for sputum, urine, blood, pleural effusion, ascites, cerebrospinal fluid and wound secretions and other body fluid samples. And the results showed that Klebsiella pneumoniae was positive, including demographic data, underlying disease status, drug sensitivity test, infection-related indicators, life support, prognostic indicators.

ELIGIBILITY:
Inclusion Criteria:

* Adult whose body fluid were sampled during ICU stay and Klebsiella pneumoniae was detected, followed by drug sensitivity test (including reporting the test results after the patient was transferred out of ICU or died).

Exclusion Criteria:

* Age were less than 18 years old;
* Patients stayed in ICU was less than 48 hours.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult whose body fluid were sampled during ICU stay and Klebsiella pneumoniae was detected, followed by drug sensitivity test.
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
prognostic indicators | 30 day
  30-day survival rate
ICU stays | about a mouth
  the length that patients stay in ICU

IPD SHARING:
Plan to Share IPD: No